CLINICAL TRIAL: NCT03976687
Title: A Phase 1b, Open-label Multiple Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of FXR Agonist/Modulator EYP001a in Healthy Volunteers and Nonalcoholic Steatohepatitis Patients
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of EYP001a in Healthy Volunteers and Nonalcoholic Steatohepatitis Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Enyo Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EYP001-107
Record Dates: First submitted 2019-06-04; First posted 2019-06-06 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: NASH - Nonalcoholic Steatohepatitis; Healthy
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 1: EYP001a Dose A (Experimental): Dose A once daily morning dose
  Interventions: Drug: EYP001a
- 2: EYP001a Dose B (Experimental): Dose B once daily morning dose
  Interventions: Drug: EYP001a
- 3: EYP001a Dose C (Experimental): Dose C twice daily - first dose morning dose and second dose 3 hours post first dose
  Interventions: Drug: EYP001a

INTERVENTIONS:
Drug: EYP001a — Oral tablets

SUMMARY:
This is a single centre, open label, randomized, 3 treatment arms, with and without food dosing, Phase 1b pharmacology study to assess the safety, tolerability, Pharmacokinetics (PK) and Pharmacodynamics (PD) of Farnesoid X Receptor (FXR) agonist/modulator EYP001a in healthy volunteers and Nonalcoholic Steatohepatitis (NASH) patients.

DETAILED DESCRIPTION:
In total 16 participants (4 healthy volunteers and 12 NASH patients) will be enrolled and randomly assigned to one of the 3 treatment arms:

* Treatment Arm 1: Dose A once daily morning dose (n=4 NASH patients, n=4 healthy volunteers)
* Treatment Arm 2: Dose B once daily morning dose (n=4 NASH patients)
* Treatment Arm 3: Dose C twice daily - first morning dose and second dose 3 hours post first dose (n=4 NASH patients).

Subsequently, all the enrolled participants (both healthy volunteers and NASH patients) will be randomly assigned to one of the 2 parallel study Groups:

* Group A (n=8, 2 healthy volunteers and 6 NASH patients): This group will include 2 NASH patients from Treatment Arms 1, 2 and 3 and 2 healthy volunteers from Treatment Arm 1. Participants in Group A will be dosed in a fasted state on Days 2, 3, 4 and 5 followed by dosing in fed state on Days 6, 7, 8 and 9.
* Group B (n=8, 2 healthy volunteers and 6 NASH patients): This group will include 2 NASH patients from Treatment Arms 1, 2 and 3 and 2 healthy volunteers from Treatment Arm 1. Participants in Group B will be dosed in a fed state on Days 2, 3, 4 and 5 followed by dosing in fasted state on Days 6, 7, 8 and 9.

The maximum total engagement duration for eligible participants in this study is up to 76 days: 60 days screening, 1-day admission visit and 8 days dosing period (in-patient in clinical trial unit) and 7 days follow-up.

The participants who are eligible for enrolment will be admitted to the Clinical Trial Unit on Day 1. The participants will receive EYP001a at the study site by trained personnel per the schedule of dosing for the study from Day 2 to Day 9 in fed/fasted state depending upon the study group. Participants will be discharged on the morning (8:00 AM) of Day 10 after collection of last PK and PD blood samples. Participants will return to the Clinical Trial Unit on Day 16 for the follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

1. Have given voluntary written informed consent;
2. Male/female participants aged 18 years to 75 years with a Body Mass Index (BMI) ≥ 25 kg/m² and ≤ 45 kg/m² at screening.
3. A female participant is eligible to participate in this study if:

   1. She is of non-childbearing potential (defined as females with a documented tubal ligation, bilateral oophorectomy or hysterectomy) or postmenopausal (defined as 12 months of spontaneous amenorrhea and follicle stimulating hormone level within the laboratory's reference range for postmenopausal females). A post-menopausal female receiving hormone replacement therapy (HRT) other than hormone replacement patches who is willing to discontinue hormone therapy 28 days before study drug dosing and agrees to remain off hormone replacement therapy for the duration of the study may be eligible for study participation. A post-menopausal female using Hormone Replacement patches who is willing to discontinue the patch 48 hours before Check in on Day -1 and until the completion of her End of Study visit is eligible for study participation.
   2. She is of childbearing potential and is non-pregnant or non-lactating and willing to use adequate contraception from screening until 3 months after the End of Study visit. Adequate contraception is defined as a progesterone only intra uterine device combined with at least 1 of the following forms of contraception: a diaphragm or cervical cap, or a condom. Also, total abstinence in accordance with the lifestyle of the participant is acceptable.
   3. She is of childbearing potential and is non-pregnant or non-lactating and taking the combined oral contraceptive pill and willing to discontinue the combined oral contraceptive pill 7 days prior to check in on Day -1 and until the completion of her End of Study visit and use adequate contraception from the day of cessation. Adequate contraception is defined as a diaphragm or cervical cap together with a condom. Also, total abstinence in accordance with the lifestyle of the participant is acceptable.
4. Have Alanine Aminotransferase (ALT) >1.5 upper limit of normal (ULN) during screening period.
5. Fibroscan® Vibration-Controlled Transient Elastography (VTCE) liver stiffness (liver stiffness measure (LSM) for >8.5 kPa) and steatosis (Controlled Attenuation Parameter (CAP) ≥250 decibels per meter (dB/m)).
6. Normal liver function at screening for alkaline phosphatase (ALP), Total Bilirubin (TBL), conjugated Bilirubin, platelets, International normalized ratio (INR).

Nota Bene: Criteria 4 and 5 do not apply to healthy volunteers.

Exclusion Criteria:

1. Employee of a contract research organization (CRO) participating in this study or the Sponsor.
2. Patients with known non-NASH chronic liver disease (alcohol, autoimmune, Human Immunodeficiency Virus (HIV), hepatitis B virus (HBV), active hepatitis C virus (HCV)).
3. Female with childbearing potential if no dual safe anti-contraception method can be provided.
4. Renal impairment (participants with an estimated glomerular filtration rate (eGFR) computed from the Modification of Diet in Renal Disease (MDRD) formula of < 60ml/min/1.73m² are excluded). Note: participants with mild renal impairment (eGFR >60 ml/min and ≤90 ml/min) are eligible.
5. Has clinically relevant immunosuppression from, but not limited to immunodeficiency conditions such as common variable hypogammaglobulinemia.
6. Has any known pre-existing medical or psychiatric condition that could interfere with the participant's ability to provide informed consent or participate in study conduct, or that may confound study findings.
7. Has a history of clinically significant gastrointestinal (GI) disease, especially peptic ulcerations, GI bleeding, ulcerative colitis, Crohn's disease or Inflammatory Bowel Syndrome, renal, hepatic, neurologic, hematologic, endocrine, oncologic, pulmonary, immunologic, or cardiovascular disease or any other condition which, in the opinion of the investigator, would jeopardize the safety of the participant or impact the validity of the study results.
8. Has participated in any drug study within 60 days prior to the first drug administration in the current study.
9. Has had major surgery within 30 days prior to the first drug administration.
10. Concomitant use of not listed drugs after discussion with Sponsor not admitted.
11. Has a history of relevant drug and/or food allergies

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-06-11 (Actual); Primary Completion 2020-05-25 (Actual); Study Completion 2020-05-25 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of EYP001a | Day 2 through day 9
Time to reach maximum concentration (Tmax) after EYP001a administration | Day 2 through day 9
Area under the concentration-time curve (AUC) from time 0 to last measurable concentration (AUC0-10h and AUClast) of EYP001a | Day 2 through day 9
Area under the concentration-time curve (AUC) and Maximum plasma concentration (Cmax) ratios | Day 2 through day 9
Type and frequencies of Adverse events | Day 1 through day 16

SECONDARY OUTCOMES:
Bile acid precursor : C4 (7αhydroxy-4-cholesten-3-one) | Day 2 through day 9
  pg/mL (picogram per milliliter). These will be measured in plasma samples using a validated method
Bile acid precursor : Fibroblast growth factor 19 (FGF19) | Day 2 through day 9
  mg/mL (milligram per milliliter). These will be measured in plasma samples using a validated method
Total Bile acids (secondary and primary) | Day 1 through day 9
  These will be measured in plasma samples using a validated method

CONTACTS AND LOCATIONS:
Locations (1):
- ENYO Pharma clinical site, Randwick, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No